CLINICAL TRIAL: NCT02087553
Title: Harmful Effects of Red Blood Cell Transfusions Are Mediated by Iron: Pediatric ICU Aim
Brief Title: PICU Transfusion Study: Harmful Effects of Red Blood Cell Transfusions
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Eldad Arie Hod, Associate Professor of Pathology and Cell Biology, Dept of Pathology&Cell Biology, Columbia University
Other Study IDs: AAAM5050; R01HL115557 (NIH)
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Iron, Abnormal Blood Level
Keywords: Blood Transfusion; Iron; Packed Red Blood Cells; PRBC; NTBI
MeSH Terms: interventions — Erythrocyte Transfusion; Sodium Chloride; Albumins

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples both pre- and post-transfusion samples of the transfusate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Transfused pediatric patients: Children who might receive packed red blood cell (PRBC) transfusion will be enrolled after obtaining consent from their parents/legal guardians and assent from the patient, if possible. Transfusion of red blood cells will be done according to standard of care.
  Interventions: Biological: Transfusion of red blood cells
- Saline/Albumin infusion: Children who might receive albumin or saline for volume resuscitation will be enrolled after obtaining consent from their parents/legal guardians and assent from the patient, if possible. Infusion will be done according to standard of care.
  Interventions: Biological: Infusion of albumin/saline

INTERVENTIONS:
Biological: Transfusion of red blood cells — (non-experimental) PRBC transfusion
  Other Names: Packed Red Blood Cells (PRBCs)
  Groups: Transfused pediatric patients
Biological: Infusion of albumin/saline — (non-experimental) albumin/saline infusion
  Other Names: Albumin/Saline
  Groups: Saline/Albumin infusion

SUMMARY:
The investigators hypothesize that the storage-damaged red cells are responsible for some of the adverse effects of transfusion. In this observational study, the investigators will measure various laboratory parameters both before and after transfusion in a pediatric intensive care unit to determine at what duration of storage is there laboratory evidence of refrigerator storage damage.

The investigators hypothesize that increasing storage time of packed red blood cells (PRBCs) transfused will be associated with increasing non-transferrin-bound iron (NTBI), pro-inﬂammatory cytokine concentrations, and enhanced microbial growth in vitro in pediatric patients.

DETAILED DESCRIPTION:
Transfusions of red blood cells (RBCs) stored for longer durations are associated with adverse effects in hospitalized patients. During storage, RBCs undergo cumulative changes that reduce their survival in vivo, and have been associated with impairment in oxygen transport and adverse outcomes. Transfusion of older RBCs results in increased NTBI levels in healthy adults, and elevated NTBI levels have been associated with increased morbidity and mortality in hospitalized patients. Transfusion of PRBCs has also been associated with up-regulation of inﬂammatory cytokines. Pediatric patients are exposed to PRBC transfusions; however, this patient population has not been previously studied for these outcomes.

According to current practice guidelines, PRBCs are stored in the blood bank up to 42 days prior to transfusion. In this study, blood sample will be collected from pediatric ICU patients prior to every PRBC transfusion and again 2-6 hours post-transfusion to determine iron parameters, inﬂammatory marker concentrations, and growth of microbial pathogens in vitro.

The investigators hopes to further the understanding of the effects of blood storage on outcome in children, thereby making transfusion safer and more effective.

ELIGIBILITY:
Inclusion Criteria:

* Less than 21 years of age;
* Greater than 5kg weight;
* Parents or legal guardian have signed informed consent;
* Will be receiving transfusion of packed, leukoreduced RBCs stored in an additive saline (AS) solution (standard practice).

Exclusion Criteria:

* Patients have undergone transfusion of platelets or fresh frozen plasma 4 hours before or will receive these products after transfusion of the RBC unit;
* Transfusion of RBC from more than one donor at the test transfusion event.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hospitalized pediatric patients admitted to the Columbia University Medical Center's Pediatric ICU
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Non-transferrin-bound iron level | Up to 12-hours post-transfusion
  Circulating non-transferrin-bound iron level post-transfusion (taken between 2-6 hours post-transfusion and 8-12 hours post-transfusion) vs the pre-transfusion level.

SECONDARY OUTCOMES:
Hepcidin level | Up to 12-hours post-transfusion
Level of C-Reactive Protein (CRP) | Up to 12 hours post-transfusion
Level of Monocyte Chemoattractant Protein (MCP)-1 | Up to 12 hours post-transfusion
Level of Interleukin (IL)-6 | Up to 12 hours post-transfusion

CONTACTS AND LOCATIONS:
Overall Officials: Eldad A Hod, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] L'Acqua C, Bandyopadhyay S, Francis RO, McMahon DJ, Nellis M, Sheth S, Kernie SG, Brittenham GM, Spitalnik SL, Hod EA. Red blood cell transfusion is associated with increased hemolysis and an acute phase response in a subset of critically ill children. Am J Hematol. 2015 Oct;90(10):915-20. doi: 10.1002/ajh.24119. PMID 26183122